CLINICAL TRIAL: NCT00004393
Title: Phase II Double Blind Placebo Controlled Trial of Risperidone in Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Yale University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199/12217; YALESM-7764
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Tourette Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
OBJECTIVES: I. Conduct a randomized, double blind, placebo controlled, parallel study of the atypical neuroleptic risperidone (RIS) in the treatment of children and adults with moderate to severe Tourette Syndrome.

II. Evaluate further the safety of RIS in this population.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled study. Initially, all patients receive placebo capsules twice daily in a single blind fashion during the first 2 weeks of study.

Then, patients are randomized to receive either risperidone (RIS) or placebo for 8 weeks. The dose of RIS is increased weekly over the first 4 weeks of treatment, as tolerated.

Patients continue RIS for 4 additional weeks at the dose prescribed during week 4.

All patients receive diagnostic evaluations at the beginning and end of the 2 week initial single blind phase, and at the end of weeks 2, 4, 6, and 8 of the active treatment phase.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

DSM-IV diagnosis of Tourette Syndrome (TS)

Tic symptoms greater than 3 (moderate or worse) on the Global Clinical Impression Scale for TS

--Prior/Concurrent Therapy--

No concurrent use of other medications during study

A minimum of 4 weeks since prior use of other medications and 8 weeks for neuroleptics or fluoxetine

--Patient Characteristics--

Hepatic: No hepatic disease

Renal: No renal disease

Cardiovascular:

* No heart disease
* No hypertension

Pulmonary: No pulmonary disease

Other:

* Not pregnant
* IQ at least 70 required
* No other movement disorder allowed, such as tardive dyskinesia
* No major depression
* No pervasive developmental disorder
* No autism or psychotic disorder based on DSM-IV
* No alcohol or substance abuse
* No hypersensitivity to risperidone
* All subjects must be in good health

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 1997-07; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S. Peterson, Study Chair — Yale University